CLINICAL TRIAL: NCT02950350
Title: Clinical Trial of Laparoscopic Pelvic and Para-aortic Lymphadenectomy and Uterine Blood Vessel Blocking for Precision Diagnosis and Treatment in Advanced Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Guo Xiaoqing
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Cervical Cancer, Stage IIB; Cervical Cancer Stage IIIA; Cervical Cancer Stage IIIB; Cervical Cancer, Stage IVA
Keywords: Cervical cancer; Precision medicine; Individualized treatment; Surgical staging
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- radiation and chemotherapy: The patients will receive radiation and chemotherapy
- removal of pelvic lymph nodes and abdominal aorta lymph nodes: The patients will receive removal of pelvic lymph nodes and abdominal aorta lymph nodes ,and receive concurrent radiation and chemotherapy

SUMMARY:
Cervical cancer is the most common reproductive malignancy in developing country. Due to local invasion, radical hysterectomy cannot be performed in advanced cervical cancer (FIGO IIB - IVA) , so that radiation combined with chemoradiation (RCTX) is a traditional treatment nowadays. Lack of precise treatment strategies, recurrent ratesand metastasisis high ,and the 5-year survival rate is less than 50%. Therefore, it needs to explore a new strategy for improving the prognosis of advanced cervical cancer.

The prognosis of cervical cancer is closely related to its stages ,while the current FIGO clinical stage is too subjective , for example different gynecologic oncologists may give different diagnosis to the same patient. MRI, CT, PET/CT imaging examinations are commonly used as a referrence for clinical staging, but the sensitivity and specificity are not satisfied. In addition, lymph node metastasis significantly impacts the prognosis of cervical cancer . However, the lymph node invasion is not in current staging criteria.

Precision treatment after surgical staging is recommended by NCCN recently .Surgical staging in patients with advancedcervical cancer is safe and does not delay primary RCTX in few randomized study.Whether overall survival benefit the long-term clinical follow-up surgical staging is unknown.Blocking bilateral uterine artery can effectively reduce the tumor size and increase the operability , which has been conformed in locally advanced cervical cancer. Furthermore, ovarian dysfunction caused by RCTX could be avoided by ovarian transposition via surgical staging .

Based on this, we suggesta new surgical stagingfor patients with advanced cervical cancer , which includinglaparoscopic pelvic and para-aortic lymphadenectomy , uterine blood vessel blocking and ovarian transportation, in order to perform individualized postoperative RCTX, reduce tumor load , preserve ovarian function and improve life quality.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis: squamous carcinoma, adenocarcinoma, adenosquamous carcinoma
* The pathological staging:IIB,IIIA,IIIB,IVA

Exclusion Criteria:

* Underwent surgery or radiation and chemotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from Dec 2016 until Dec 2018 in Shanghai First Maternity and Infant Hospital, Tongji University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate | 5 years after treatment

SECONDARY OUTCOMES:
The transfer rate | 5 years after treatment
mortality | 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqing Guo, PHD, Principal Investigator — Shanghai First Maternity and Infant Hospital

IPD SHARING:
Plan to Share IPD: Undecided
we need get the patients' agreement to share data.